CLINICAL TRIAL: NCT00073749
Title: A Phase 1 Study Of Cmc-544 Administered As A Single Agent In Subjects With B-cell Non- Hodgkin's Lymphoma
Brief Title: Study Evaluating CMC-544 In B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 3129K1-100; B1931002 (Other: Alias Study Number)
Record Dates: First submitted 2003-12-04; First posted 2003-12-05 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Lymphoma, B-Cell
Keywords: B-Cell; Non-Hodgkin's; Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inotuzumab ozogamicin (Experimental): Inotuzumab ozogamicin, iv, dose escalation and expanded cohort at 1.8mg/m2
  Interventions: Drug: Inotuzumab ozogamicin [CMC-544]

INTERVENTIONS:
Drug: Inotuzumab ozogamicin [CMC-544] — CMC-544, IV, dose escalation trial

SUMMARY:
To determine the Maximum Tolerated Dose (MTD), the tolerability, and the initial safety profile of CMC-544 in subjects with B-cell Non-Hodgkin's Lymphoma (NHL).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been previously diagnosed with CD22-positive, B-cell NHL, according to WHO classification, which has progressed after at least 2 prior therapies of probable clinical benefit
* At the expanded cohort, part 2 of the study, subjects must have one of the following:
* Follicular lymphoma previously treated with at least one dose of rituximab, but have not received radioimmunotherapy
* Diffuse large B-cell lymphoma
* Age 18 years or older

Exclusion Criteria:

* Candidate for potentially curative therapies in the opinion of the investigator
* Chronic lymphocytic leukemia
* Burkitt's lymphoma, primary effusion lymphoma, and precursor B-cell lymphoblastic lymphoma

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2003-08 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (11):
  - UAB CCC Clinical Studies Unit, Birmingham, Alabama
  - University of Alabama at Birmingham Kirklin Clinic, Birmingham, Alabama
  - UAB Russell Ambulatory Pharmacy, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - M.D. Anderson Cancer Center, Houston, Texas
- Universitair Ziekenhuis Gasthuisberg, Leuven, Belgium
- France (2):
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
- Germany (4):
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet, Mainz
  - Medizinische Klinik und Poliklinik III, Klinikum der Universitat Muenchen-Grosshadern, München
  - Universitaet Muenchen Klinikum Grosshadern, München
- Spain (2):
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Clinic I Provincial, Barcelona
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- St Bartholomew's Hospital, London, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3129K1-100&StudyName=Study%20Evaluating%20CMC-544%20In%20B-Cell%20Non-Hodgkin%27s%20Lymphoma

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in 2 parts. Part 1: Dose escalation cohorts of inotuzumab ozogamicin to determine the maximum tolerated dose (MTD) included 21 days and 28 days dose administration cycles. Part 2: Expanded cohort using the MTD regimen identified in Part 1.
Groups:
- Inotuzumab Ozogamicin 0.4 mg/m^2: Dose Escalation Cohort 1: Participants with CD22-positive B-cell non-Hodgkin lymphoma (NHL) received 0.4 milligrams per square meter (mg/m^2) intravenous (IV) dose of inotuzumab ozogamicin on Day 1 of each cycle, for at least 4 cycles unless there was an evidence of disease progression or unacceptable toxicity. Each cycle was of 21 days.
- Inotuzumab Ozogamicin 0.8 mg/m^2: Dose Escalation Cohort 2: Participants with CD22-positive B-cell NHL received 0.8 mg/m^2 IV dose of inotuzumab ozogamicin on Day 1 of each cycle, for at least 4 cycles, unless there was an evidence of disease progression or unacceptable toxicity. Each cycle was of 21 days.
- Inotuzumab Ozogamicin 1.34 mg/m^2: Dose Escalation Cohort 3: Participants with CD22-positive B-cell NHL received 1.34 mg/m^2 IV dose of inotuzumab ozogamicin on Day 1 of each cycle, for at least 4 cycles, unless there was evidence of disease progression or unacceptable toxicity. Each cycle was of 21 days.
- Inotuzumab Ozogamicin 1.8 mg/m^2: Dose Escalation Cohort 4: Participants with CD22-positive B-cell NHL received 1.8 mg/m^2 IV dose of inotuzumab ozogamicin on Day 1 of each cycle, for at least 4 cycles, unless there was evidence of disease progression or unacceptable toxicity. Each cycle was of 21 days.
- Inotuzumab Ozogamicin 2.4 mg/m^2: Dose Escalation Cohort 5: Participants with CD22-positive B-cell NHL received 2.4 mg/m^2 IV dose of inotuzumab ozogamicin on Day 1 of each cycle, for at least 4 cycles, unless there was evidence of disease progression or unacceptable toxicity. Each cycle was of 21 days.
- Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in Cohort; Inotuzumab Ozogamicin 1.8 mg/m^2: Expanded Cohort: Participants with CD22-positive B-cell NHL received 1.8 mg/m^2 IV dose of inotuzumab ozogamicin on Day 1 of each cycle, for at least 4 cycles, unless there was evidence of disease progression or unacceptable toxicity. Each cycle was of 28 days.
Period: Overall Study
Arm/Group | Inotuzumab Ozogamicin 0.4 mg/m^2: Dose Escalation Cohort 1 | Inotuzumab Ozogamicin 0.8 mg/m^2: Dose Escalation Cohort 2 | Inotuzumab Ozogamicin 1.34 mg/m^2: Dose Escalation Cohort 3 | Inotuzumab Ozogamicin 1.8 mg/m^2: Dose Escalation Cohort 4 | Inotuzumab Ozogamicin 2.4 mg/m^2: Dose Escalation Cohort 5 | Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in Cohort | Inotuzumab Ozogamicin 1.8 mg/m^2: Expanded Cohort
Started | 2 | 5 | 11 | 6 | 6 | 6 | 43
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not Completed | 2 | 5 | 11 | 6 | 6 | 6 | 40
Not completed — Disease Progression | 2 | 0 | 3 | 2 | 3 | 1 | 3
Not completed — Death | 0 | 1 | 1 | 0 | 0 | 0 | 29
Not completed — Adverse Event | 0 | 3 | 6 | 4 | 2 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1 | 0 | 2
Not completed — Discontinuation of Study by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population included all participants who received at least 1 dose of inotuzumab ozogamicin.
Groups:
- Total: Total of all reporting groups
Arm/Group | Inotuzumab Ozogamicin 0.4 mg/m^2: Dose Escalation Cohort 1 | Inotuzumab Ozogamicin 0.8 mg/m^2: Dose Escalation Cohort 2 | Inotuzumab Ozogamicin 1.34 mg/m^2: Dose Escalation Cohort 3 | Inotuzumab Ozogamicin 1.8 mg/m^2: Dose Escalation Cohort 4 | Inotuzumab Ozogamicin 2.4 mg/m^2: Dose Escalation Cohort 5 | Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in Cohort | Inotuzumab Ozogamicin 1.8 mg/m^2: Expanded Cohort | Total
Number analyzed (Participants) | 2 | 5 | 11 | 6 | 6 | 6 | 43 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.50 (13.44) | 73.80 (2.59) | 65.45 (10.56) | 56.67 (5.96) | 60.00 (12.82) | 57.17 (12.25) | 57.30 (10.91) | 59.46 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 4 | 0 | 1 | 2 | 23 | 32
  Male | 2 | 3 | 7 | 6 | 5 | 4 | 20 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent adverse events (TEAE) are defined as any new event reported after first dose of study drug up to 42 days after last dose of study drug, or any event that is worse in severity than at any time during the baseline period. AEs included both SAEs and non-serious adverse events (non-SAEs).
Time Frame: Baseline up to 42 days after last dose of study drug (up to Day 225)
Population: Safety population included all participants who received at least 1 dose of inotuzumab ozogamicin.
Measure: Number; unit: participants
Groups:
- Inotuzumab Ozogamicin: Dose Escalation Cohorts 1 to 5: Participants with CD22-positive B-cell NHL received 0.4 or 0.8 or 1.34 or 1.8 or 2.4 mg/m^2 intravenous (IV) dose of inotuzumab ozogamicin on Day 1 of each cycle, for at least 4 cycles unless there was an evidence of disease progression or unacceptable toxicity. Each cycle was of 21 days.
- Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in + Expanded Cohorts: Participants with CD22-positive B-cell NHL received 1.8 mg/m^2 IV dose of inotuzumab ozogamicin on Day 1 of each cycle, for at least 4 cycles, unless there was evidence of disease progression or unacceptable toxicity. Each cycle was of 28 days.
Arm/Group | Inotuzumab Ozogamicin: Dose Escalation Cohorts 1 to 5 | Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in + Expanded Cohorts
Number analyzed (Participants) | 30 | 49
participants
  AEs | 29 | 49
  SAEs | 11 | 15

2. Primary Outcome: Number of Participants With Grade 3 or Higher Grades Treatment-Emergent Adverse Events (TEAEs) Based on Severity
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AE severity was defined to be the maximum toxicity grade of the treatment-emergent adverse events (TEAEs) experienced by the participants during the study. AE was assessed according to severity; Grade 1 (mild AE), Grade 2 (moderate AE), Grade 3 (severe AE), Grade 4 (life-threatening or disabling AE), Grade 5 (death related to AE). Participants with Grade 3 or higher grades TEAEs were reported.
Time Frame: Baseline up to 42 days after last dose of study drug (up to Day 225)
Population: Safety population included all participants who received at least 1 dose of inotuzumab ozogamicin.
Measure: Number; unit: participants
Arm/Group | Inotuzumab Ozogamicin: Dose Escalation Cohorts 1 to 5 | Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in + Expanded Cohorts
Number analyzed (Participants) | 30 | 49
participants | 24 | 42

3. Primary Outcome: Maximum Tolerated Dose (MTD): Part 1 (Dose Escalation Cohorts)
Description: MTD was defined as highest dose level for which no more than 1 participant in a dose cohort experienced dose limiting toxicity (DLT). DLT was defined as any of the following events occurring during the first 21 days (or 28 days for participants treated every 4 weeks) days of study medication and considered at least possibly-related to study medication: any grade 3 or 4 non-hematologic toxicity except grade 3 alopecia, nausea, or vomiting, any grade 4 febrile neutropenia, any grade 4 thrombocytopenia or any bleeding episode requiring platelet transfusion, any grade 4 absolute neutrophil count (for a duration of greater than or equal to [>=] 7 days), delayed recovery (less than or equal to [<=] grade 1 or baseline) from a toxicity that delays the initiation of the next dose by more than 2 weeks.
Time Frame: Baseline up to Day 28
Population: Safety population included all participants who received at least 1 dose of inotuzumab ozogamicin. This outcome measure was not planned to be analyzed in Part 2 of the study.
Measure: Number; unit: milligram per meter square (mg/m^2)
Groups:
- Inotuzumab Ozogamicin: Dose Escalation Cohorts 1 to 5: Participants with CD22-positive B-cell NHL received either 0.4, 0.8, 1.34, 1.8 or 2.4 mg/m^2 IV dose of inotuzumab ozogamicin on Day 1 of each cycle, for at least 4 cycles unless there was an evidence of disease progression or unacceptable toxicity. Each cycle was of 21 days.
Arm/Group | Inotuzumab Ozogamicin: Dose Escalation Cohorts 1 to 5
Number analyzed (Participants) | 30
milligram per meter square (mg/m^2) | 1.8

4. Primary Outcome: Number of Participants With Dose-limiting Toxicity (DLT)
Description: DLT was classified as per National Cancer Institute common terminology criteria for adverse events (NCI CTCAE) version 3.0 and defined as any of the following events occurring during the first 21 days (or 28 days for participants treated every 4 weeks) days of study medication and considered at least possibly-related to study medication: any grade 3 or 4 non-hematologic toxicity except grade 3 alopecia, nausea, or vomiting, any grade 4 febrile neutropenia, any grade 4 thrombocytopenia or any bleeding episode requiring platelet transfusion, any grade 4 absolute neutrophil count (for a duration of greater than or equal to [>=] 7 days), delayed recovery (less than or equal to [<=] grade 1 or baseline) from a toxicity that delays the initiation of the next dose by more than 14 days.
Time Frame: Baseline up to Day 28
Population: Safety population included all participants who received at least 1 dose of inotuzumab ozogamicin. Here number of participant analyzed (N) signifies participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Inotuzumab Ozogamicin 0.4 mg/m^2: Dose Escalation Cohort 1 | Inotuzumab Ozogamicin 0.8 mg/m^2: Dose Escalation Cohort 2 | Inotuzumab Ozogamicin 1.34 mg/m^2: Dose Escalation Cohort 3 | Inotuzumab Ozogamicin 1.8 mg/m^2: Dose Escalation Cohort 4 | Inotuzumab Ozogamicin 2.4 mg/m^2: Dose Escalation Cohort 5 | Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in + Expanded Cohorts
Number analyzed (Participants) | 2 | 5 | 11 | 6 | 6 | 6
participants | 0 | 0 | 2 | 1 | 2 | 0

5. Secondary Outcome: Progression-Free Survival (PFS): Evaluable Population- Part 2 (Lead-in + Expanded Cohorts)
Description: PFS was based on Kaplan-Meier estimates. PFS was defined as the time interval from the first dose of study medication until the first date on which relapsed disease, or progression (as per the International Response Criteria for Non-Hodgkin Lymphoma) or death, was documented, censored at the last tumor evaluation date. This outcome measure was analyzed in participants with follicular lymphoma or diffuse large B-cell lymphoma.
Time Frame: Baseline, every 8 weeks up to Year 1, then every 12 weeks up to Year 2, and then every 6 months until tumor progression or death (up to Year 5)
Population: Evaluable population: All participants who received at least 2 doses of study drug, had baseline tumor computed tomography (CT) scan, and at least 1 post-baseline tumor assessment for anti-cancer clinical activity. Here 'N' represents number of participants evaluable for this outcome measure. This was not planned to be analyzed in Part 1 of study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in + Expanded Cohorts
Number analyzed (Participants) | 35
days
  With Diffuse Lymphoma: number analyzed (Participants) | 16
  With Diffuse Lymphoma | 103 [52 to 135]
  With Follicular Lymphoma: number analyzed (Participants) | 19
  With Follicular Lymphoma | 311 [211 to 569]

6. Secondary Outcome: Progression-Free Survival (PFS): Intent-to-treat Population-Part 2 (Lead-in + Expanded Cohorts)
Description: PFS was based on Kaplan-Meier estimates. PFS was defined as the time interval from the first dose of study medication until the first date on which relapsed disease, or progression (as per International Response Criteria for Non-Hodgkin Lymphoma) or death, was documented, censored at the last tumor evaluation date. This outcome measure was analyzed in participants with follicular lymphoma or diffuse large B-cell lymphoma.
Time Frame: as for outcome 5
Population: Intent-to-treat (ITT) population included all enrolled participants. Here 'N' represents number of participants evaluable for this outcome measure. This outcome measure was not planned to be analyzed in Part 1 of the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in + Expanded Cohorts
Number analyzed (Participants) | 48
days
  With Diffuse Lymphoma: number analyzed (Participants) | 26
  With Diffuse Lymphoma | 49.5 [29 to 100]
  With Follicular Lymphoma: number analyzed (Participants) | 22
  With Follicular Lymphoma | 254 [182 to 386]

7. Secondary Outcome: Overall Survival (OS): Evaluable Population- Part 2 (Lead-in + Expanded Cohorts)
Description: OS was based on Kaplan-Meier method. Survival was defined as the time period from the first dose of study drug until the date of death, censored at the participant's last contact date. This outcome measure was analyzed in participants with follicular lymphoma or diffuse large B-cell lymphoma.
Time Frame: Baseline up to Year 5
Population: Evaluable population: All participants who received at least 2 doses of study drug, had baseline tumor CT scan, and at least 1 post-baseline tumor assessment for anti-cancer clinical activity. Here 'N' represents number of participants evaluable for this outcome measure. This outcome measure was not planned to be analyzed in Part 1 of study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in + Expanded Cohorts
Number analyzed (Participants) | 35
days
  With Diffuse Lymphoma: number analyzed (Participants) | 16
  With Diffuse Lymphoma | 274 [169 to 519]
  With Follicular Lymphoma: number analyzed (Participants) | 19
  With Follicular Lymphoma | NA [NA to NA] — Data not collected since median overall survival was not reached for the participants with follicular lymphoma.

8. Secondary Outcome: Overall Survival (OS): Intent-to-treat Population: Part 2 (Lead-in + Expanded Cohorts)
Description: Interval OS was based on Kaplan-Meier method. Survival was defined as the time period from the first dose of study drug until the date of death, censored at the participant's last contact date. This outcome measure was analyzed in participants with follicular lymphoma or diffuse large B-cell lymphoma.
Time Frame: Baseline up to Year 5
Population: ITT population included all enrolled participants. Here 'N' signifies number of participants evaluable for this outcome measure. This outcome measure was not planned to be analyzed in Part 1 of the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in + Expanded Cohorts
Number analyzed (Participants) | 48
days
  With Diffuse Lymphoma: number analyzed (Participants) | 26
  With Diffuse Lymphoma | 194 [128 to 363]
  With Follicular Lymphoma: number analyzed (Participants) | 22
  With Follicular Lymphoma | 1147 [523 to NA] — Data not collected since upper limit for overall survival was not reached for participants with follicular lymphoma.

9. Secondary Outcome: Number of Participants With Best Overall Response (BOR): Part 2 (Expanded Cohorts)
Description: Participants with BOR=with complete response(CR),unconfirmed CR(CRu) or partial response (PR) as per International Response Criteria for NHL. CR: Total disappearance of all detectable clinical,radiographic sign of disease/related symptoms,normalization biochemical abnormalities related to NHL;if enlarged before therapy all lymph nodes,nodal masses,other organs regressed to normal size and spleen regressed in size,undetectable on physical exam,clear bone marrow infiltrate. CRu: CR but allows for residual lymph node mass >1.5 cm in greatest transverse diameter and all individual nodes previously merged were regressed by >75% in product diameters and indeterminate bone marrow. PR:>=50% decrease in sum of products of greatest diameters(SPD) of 6 largest dominant nodes/nodal masses,no increase in size of other nodes/spleen/liver, 50% decrease in SPD of splenic,hepatic nodules,involvement of other organs considered assessable,not measurable disease with exception of splenic,hepatic nodules.
Time Frame: as for outcome 5
Population: Evaluable population was analyzed. Participants with diffuse or follicular lymphoma were analyzed. This outcome measure was not planned to be analyzed in Part 1 and Part 2 (Lead-in Cohort).
Measure: Number; unit: participants
Arm/Group | Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in + Expanded Cohorts
Number analyzed (Participants) | 30
participants
  CR: With Follicular Lymphoma: number analyzed (Participants) | 15
  CR: With Follicular Lymphoma | 1
  CR: With Diffuse Lymphoma: number analyzed (Participants) | 15
  CR: With Diffuse Lymphoma | 2
  CRu: With Follicular Lymphoma: number analyzed (Participants) | 15
  CRu: With Follicular Lymphoma | 3
  CRu: With Diffuse Lymphoma: number analyzed (Participants) | 15
  CRu: With Diffuse Lymphoma | 0
  PR: With Follicular Lymphoma: number analyzed (Participants) | 15
  PR: With Follicular Lymphoma | 8
  PR: With Diffuse Lymphoma: number analyzed (Participants) | 15
  PR: With Diffuse Lymphoma | 5

10. Secondary Outcome: Duration of Overall Response (DoR): Part 2 (Lead-in + Expanded Cohorts)
Description: Duration of overall response was defined as the time from the date that measurement criteria were met for CR, CRu, or PR (whichever status was recorded first) until the first date that relapsed disease was objectively documented as per International Response Criteria for NHL, taking as reference for relapsed disease the smallest measurements recorded since the treatment started. This outcome measure was analyzed in participants with follicular lymphoma or diffuse large B-cell lymphoma.
Time Frame: as for outcome 5
Population: Evaluable population was analyzed. DoR included evaluable participants who achieved CR, CRu, or PR. Here 'N' signifies number of participants evaluable for this outcome measure. This outcome measure was not planned to be analyzed in Part 1 of the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in + Expanded Cohorts
Number analyzed (Participants) | 22
days
  With Diffuse Lymphoma: number analyzed (Participants) | 7
  With Diffuse Lymphoma | 80.00 [42.00 to 1637]
  With Follicular Lymphoma: number analyzed (Participants) | 15
  With Follicular Lymphoma | 233.0 [130.0 to 520.0]

11. Secondary Outcome: Time-to-Tumor Progression: Part 2 (Expanded Cohorts)
Description: Time to tumor progression was defined as the interval from the start of the treatment until the first date on which relapsed disease or progression is documented, censored at the last disease assessment. This outcome measure was analyzed in participants with follicular lymphoma or diffuse large B-cell lymphoma.
Time Frame: as for outcome 5
Population: Evaluable population was analyzed. Here "N" signifies number of participants evaluable for this outcome measure. This outcome measure was not planned to be analyzed in Part 1 and Part 2 (Lead-in Cohort) of the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in + Expanded Cohorts
Number analyzed (Participants) | 30
days
  With Diffuse Lymphoma: number analyzed (Participants) | 15
  With Diffuse Lymphoma | 105 [55 to NA] — Data not collected since upper limit for time to tumor progression was not reached.
  With Follicular Lymphoma: number analyzed (Participants) | 15
  With Follicular Lymphoma | 339 [189 to NA] — Data not collected since upper limit for time to tumor progression was not reached.

12. Other Pre Specified Outcome: Percentage of Participants With Objective Response- Evaluable Population: Part 2 (Lead-in + Expanded Cohorts)
Description: Participants (having follicular or diffuse lymphoma) with objective response based assessment of CR, CRu or PR as per International Response Criteria for NHL. CR: Total disappearance of all detectable clinical, radiographic sign of disease/related symptoms, normalization biochemical abnormalities related to NHL; if enlarged before therapy all lymph nodes, nodal masses, other organs regressed to normal size and spleen regressed in size, undetectable on physical exam, clear bone marrow infiltrate. CRu: CR but allows for residual lymph node mass >1.5 cm in greatest transverse diameter and all individual nodes previously merged were regressed by >75% in product diameters and indeterminate bone marrow. PR: >=50% decrease in SPD of 6 largest dominant nodes or nodal masses, no increase in size of other nodes, spleen or liver, 50% decrease in SPD of splenic, hepatic nodules, involvement of other organs considered assessable, not measurable disease with exception of splenic, hepatic nodules.
Time Frame: Baseline up to 42 days after last dose (Day 225)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in + Expanded Cohorts
Number analyzed (Participants) | 35
percentage of participants
  With Diffuse Lymphoma: number analyzed (Participants) | 16
  With Diffuse Lymphoma | 25 [7.27 to 52.38]
  With Follicular Lymphoma: number analyzed (Participants) | 19
  With Follicular Lymphoma | 73.68 [48.80 to 90.85]

13. Other Pre Specified Outcome: Percentage of Participants With Objective Response- Intent-to-treat Population: Part 2 (Lead in+ Expanded Cohorts)
Description: as for outcome 12
Time Frame: Baseline up to 42 days after last dose of study drug (Day 225)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in + Expanded Cohorts
Number analyzed (Participants) | 48
percentage of particpants
  With Diffuse Lymphoma: number analyzed (Participants) | 26
  With Diffuse Lymphoma | 15.38 [4.36 to 34.87]
  With Follicular Lymphoma: number analyzed (Participants) | 22
  With Follicular Lymphoma | 68.12 [45.13 to 86.14]

ADVERSE EVENTS:
Time Frame: Treatment-emergent events: Baseline up to 42 days after last dose of study drug (up to Day 225)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as non-serious in another subject, or one subject may have experienced both a serious and non-serious event during the study.
Arm/Group | Inotuzumab Ozogamicin 0.4 mg/m^2: Dose Escalation Cohort 1 | Inotuzumab Ozogamicin 0.8 mg/m^2: Dose Escalation Cohort 2 | Inotuzumab Ozogamicin 1.34 mg/m^2: Dose Escalation Cohort 3 | Inotuzumab Ozogamicin 1.8 mg/m^2: Dose Escalation Cohort 4 | Inotuzumab Ozogamicin 2.4 mg/m^2: Dose Escalation Cohort 5 | Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in Cohort | Inotuzumab Ozogamicin 1.8 mg/m^2: Expanded Cohort
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/5 | 3/11 | 3/6 | 4/6 | 0/6 | 15/43
Other Adverse Events (participants affected / at risk) | 1/2 | 5/5 | 11/11 | 6/6 | 6/6 | 6/6 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inotuzumab Ozogamicin 0.4 mg/m^2: Dose Escalation Cohort 1 (N=2) | Inotuzumab Ozogamicin 0.8 mg/m^2: Dose Escalation Cohort 2 (N=5) | Inotuzumab Ozogamicin 1.34 mg/m^2: Dose Escalation Cohort 3 (N=11) | Inotuzumab Ozogamicin 1.8 mg/m^2: Dose Escalation Cohort 4 (N=6) | Inotuzumab Ozogamicin 2.4 mg/m^2: Dose Escalation Cohort 5 (N=6) | Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in Cohort (N=6) | Inotuzumab Ozogamicin 1.8 mg/m^2: Expanded Cohort (N=43)
FEVER (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 3
ASTHENIA (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
ASCITES (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
SEPSIS (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
BACK PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
CELLULITIS (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
CHILLS (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
DEATH (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HERNIA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
MALAISE (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
NEUTROPENIC FEVER (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
PAIN (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
DEEP VEIN THROMBOSIS (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
SYNCOPE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
LIVER FUNCTION TESTS ABNORMAL (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
ANOREXIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
DIARRHEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
VENOOCCLUSIVE LIVER DISEASE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 2 | 0 | 3
LYMPHOMA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
BILIRUBINEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
CACHEXIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
LACTIC DEHYDROGENASE INCREASED (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
MENTAL STATUS CHANGES (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
NEUROPATHY (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
ACUTE KIDNEY FAILURE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inotuzumab Ozogamicin 0.4 mg/m^2: Dose Escalation Cohort 1 (N=2) | Inotuzumab Ozogamicin 0.8 mg/m^2: Dose Escalation Cohort 2 (N=5) | Inotuzumab Ozogamicin 1.34 mg/m^2: Dose Escalation Cohort 3 (N=11) | Inotuzumab Ozogamicin 1.8 mg/m^2: Dose Escalation Cohort 4 (N=6) | Inotuzumab Ozogamicin 2.4 mg/m^2: Dose Escalation Cohort 5 (N=6) | Inotuzumab Ozogamicin 1.8 mg/m^2: Lead-in Cohort (N=6) | Inotuzumab Ozogamicin 1.8 mg/m^2: Expanded Cohort (N=43)
ASTHENIA (General disorders) | 1 | 4 | 7 | 3 | 4 | 2 | 30
HEMORRHAGE (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
HYPOTENSION (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1
EXTRASYSTOLES (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
HYPERTENSION (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
VASODILATATION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
BUNDLE BRANCH BLOCK (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
MIGRAINE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
MYOCARDIAL ISCHEMIA (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
PALLOR (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
PERIPHERAL VASCULAR DISORDER (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
PHLEBITIS (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
POSTURAL HYPOTENSION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
SHOCK (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
SYNCOPE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
VASCULAR ANOMALY (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
VASCULAR DISORDER (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
VASCULITIS (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 3 | 6 | 4 | 2 | 4 | 20
ANOREXIA (Gastrointestinal disorders) | 0 | 2 | 3 | 1 | 3 | 3 | 12
CONSTIPATION (Gastrointestinal disorders) | 0 | 2 | 3 | 1 | 1 | 2 | 10
DIARRHEA (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 3 | 1 | 8
VOMITING (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 0 | 2 | 10
GAMMA GLUTAMYL TRANSPEPTIDASE INCREASED (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 1 | 0 | 4
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 6
DRY MOUTH (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 3
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 2
STOMATITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2
LIVER FUNCTION TESTS ABNORMAL (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2
ERUCTATION (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
FLATULENCE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
GASTROENTERITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
GUM HEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
MUCOSITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
BLOOD IN STOOL (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
CHOLELITHIASIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
FECAL INCONTINENCE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
HEPATOMEGALY (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
LIVER FATTY DEPOSIT (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
MOUTH ULCERATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
NAUSEA AND VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
ORAL MONILIASIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
PANCREAS DISORDER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
RECTAL DISORDER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 3 | 8 | 6 | 5 | 6 | 38
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1 | 3 | 2 | 3 | 4 | 21
ANEMIA (Blood and lymphatic system disorders) | 0 | 0 | 3 | 1 | 1 | 1 | 12
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 1 | 1 | 12
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 1 | 2 | 6
ECCHYMOSIS (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 3
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
FIBRINOGEN INCREASED (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
GRANULOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
INTERNATIONAL NORMALISED RATIO INCREASED (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
LYMPHOMA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
THROMBIN TIME PROLONGED (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
LYMPHOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
MEGAKARYOCYTES DECREASED (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
PETECHIAE (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
PURPURA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
RETICULOENDOTHELIAL HYPERPLASIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
SPLENOMEGALY (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
SGOT INCREASED (Metabolism and nutrition disorders) | 0 | 0 | 5 | 4 | 2 | 2 | 18
ALKALINE PHOSPHATASE INCREASED (Metabolism and nutrition disorders) | 1 | 0 | 4 | 2 | 1 | 2 | 11
SGPT INCREASED (Metabolism and nutrition disorders) | 0 | 0 | 4 | 3 | 1 | 1 | 8
BILIRUBINEMIA (Metabolism and nutrition disorders) | 0 | 0 | 3 | 1 | 1 | 0 | 11
PERIPHERAL EDEMA (Metabolism and nutrition disorders) | 0 | 2 | 3 | 0 | 0 | 0 | 10
HYPOKALEMIA (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1 | 0 | 1 | 6
LACTIC DEHYDROGENASE INCREASED (Metabolism and nutrition disorders) | 0 | 0 | 4 | 2 | 2 | 0 | 4
HYPOPROTEINEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 6
WEIGHT LOSS (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 3
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 3
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4
HYPERURICEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4
CREATININE INCREASED (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
EDEMA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
HYPERCHOLESTEREMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
HYPONATREMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
BUN INCREASED (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
HYPERCALCEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
ACIDOSIS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
CACHEXIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPERCHLOREMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPERLIPEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPOCALCEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
HYPOCHLOREMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
WEIGHT GAIN (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 1 | 0 | 0 | 6
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
MYASTHENIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
JOINT DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
MUSCLE ATROPHY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
TENDON DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 5
PARESTHESIA (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 4
INSOMNIA (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 3
ANXIETY (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 4
DEPRESSION (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1
NEUROPATHY (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
NERVOUSNESS (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
SOMNOLENCE (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
AGITATION (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
APHASIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
ATAXIA (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
CLONUS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
FACIAL PARALYSIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
HYPESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
MENTAL STATUS CHANGES (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
MYELOPATHY (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
NEUROPATHIC PAIN (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
TREMOR (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
COUGH INCREASED (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 0 | 1 | 4 | 7
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2 | 0 | 3 | 6
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 2 | 0 | 0 | 6
RHINITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 3 | 7
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 4
SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 3
UPPER RESPIRATORY INFECTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 2
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
PULMONARY PHYSICAL FINDING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
HICCUP (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
VOICE ALTERATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
ALVEOLITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
LUNG INFILTRATION NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
PLEURAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
SPUTUM INCREASED (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 3
SWEATING (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 3
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
HERPES SIMPLEX (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
HERPES ZOSTER (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
FOLLICULITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
FUNGAL DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
PRURITIC RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
SKIN BENIGN NEOPLASM (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
SKIN DISCOLORATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
URINARY TRACT INFECTION (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
ALBUMINURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
BREAST PAIN (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
CYSTITIS (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
DYSURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
HEMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OLIGURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
TESTIS DISORDER (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
URINARY FREQUENCY (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
URINARY HESITATION (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
URINE ABNORMALITY (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
FEVER (General disorders) | 0 | 0 | 2 | 3 | 3 | 4 | 17
ABDOMINAL PAIN (General disorders) | 1 | 1 | 5 | 4 | 2 | 1 | 14
HEADACHE (General disorders) | 0 | 0 | 4 | 3 | 0 | 1 | 9
BACK PAIN (General disorders) | 1 | 0 | 5 | 0 | 1 | 2 | 4
PAIN (General disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 7
CHILLS (General disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 6
LAB TEST ABNORMAL (General disorders) | 0 | 0 | 2 | 2 | 1 | 0 | 3
CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 5
INFECTION (General disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 2
ABDOMEN ENLARGED (General disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0
ACCIDENTAL INJURY (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
FLU SYNDROME (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
NECK PAIN (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1
ASCITES (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
PELVIC PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
ALLERGIC REACTION (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
FACE EDEMA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
IMMUNOGLOBULINS DECREASED (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
INJECTION SITE REACTION (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
NEOPLASM (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
RADIATION INJURY (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
CONJUNCTIVITIS (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1
ABNORMAL VISION (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
EYE DISORDER (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1
DRY EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
CATARACT SPECIFIED (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
CORNEAL LESION (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
EYE PAIN (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
TASTE PERVERSION (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 2
EAR PAIN (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
BLEPHARITIS (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
EAR DISORDER (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
KERATITIS (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
TASTE LOSS (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
REACTION UNEVALUABLE (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
ALLERGIC REACTION OTHER THAN DRUG (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
DEVICE MALFUNCTION (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.